CLINICAL TRIAL: NCT05157893
Title: Effects of Virtual Reality (VR) Based Distraction and Relaxation Therapy on Moderate and Severe Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-21-011
Record Dates: First submitted 2021-11-30; First posted 2021-12-15 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: pain; virtual reality; distraction therapy; relaxation therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR analgesic therapy (Experimental): Patients receive a single VR therapy lasting 15 min.
  Interventions: Device: Virtual reality based analgesic therapy

INTERVENTIONS:
Device: Virtual reality based analgesic therapy — The intervention is a single 15 min VR therapy. The VR therapy is consisted of VR device and software. The model of VR device used is Pico Neo 3 Pro. The software run on the VR device delivers two types of contents: 1) A 7min of computer-generated 360 video of underwater scene with therapeutic music to distract patients' attention on pain and make patients passively relax. 2) An 8min guided relaxation in which patients are transported to seaside with narrative to achieve image and breathing relaxation.

SUMMARY:
This is a prospective, single-arm, open, single-center clinical study. This study is a pilot study to explore the use of VR based distraction and relaxation therapy as an adjunctive analgesic method for Chinese patients with moderate to severe pain. After screening, patients with moderate to severe pain who meet the study inclusion criteria receive VR therapy for 15 minutes to evaluate the effectiveness and safety of VR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years old.
* Average pain intensity≥4 on a 0-10 numerical rating scale (NRS) in the past 24 hours.
* Be able to communicate in Chinese.
* Be able to read and write Chinese.
* Willing to comply with study procedures and restrictions.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Shingles on the eyes, ears, head, face, or hands.
* Trigeminal neuralgia.
* Severe vision impairment. (Patients with clear vision wearing glasses or contact lenses are allowed)
* Severe hearing impairment.
* Disease or medical condition predisposing to nausea or dizziness, such as insufficient blood supply to the brain, vestibular dysfunction, cholecystitis, etc.
* History of severe motion sickness.
* Injury to eyes, ears, face, or neck that impedes comfortable use of virtual reality.
* Injury or dysfunction of hands or upper limbs that impedes comfortable use of virtual reality.
* Diagnosis of cognitive impairment, epilepsy, dementia, migraines or other neurological diseases that may prevent the use of virtual reality.
* History of mental illness, including depression, generalized anxiety disorder, schizophrenia, etc.
* Females currently pregnant.
* Current or completion of participation within 4 weeks before screening in any interventional clinical study
* Patients whom the investigator considers not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity before and after VR therapy | 20min
  The pain intensity is measured using a 0-10 numerical rating scale (NRS) of pain. The anchors for the numerical rating scale were "Ten is the worst pain anyone could ever have and zero is no pain at all." Before the VR therapy started, the participant would be asked what his or her pain level is on the 0-10 numerical rating scale. After the 15 minute VR therapy, the participant would be asked what his or her pain level at that moment, again using the 0-10 numerical rating scale. The change in pain intensity before and after VR therapy is then obtained with the two pain level numbers subtracted.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai XINHUA Hospital, Shanghai, China